CLINICAL TRIAL: NCT06488742
Title: Efficacy of 3% Kanuka Oil Versus 1% Hydrocortisone Cream in the Treatment of Patients With Mild Atopic Dermatitis
Brief Title: The Efficacy of 3% Kanuka Oil Versus 1% Hydrocortisone Cream in Patients With Atopic Dermatitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nexgen Dermatologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KO-104
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Dermatitis, Atopic; Pruritus
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3% Kanuka Oil Cream (Experimental): 3% kanuka oil cream will be applied topically to the affected area twice a day for 28 days
  Interventions: Other: 3% kanuka oil
- 1% Hydrocortisone Cream (Active Comparator): 1% Hydrocortisone Cream will be applied topically to the affected area twice a day for 28 days
  Interventions: Other: 3% kanuka oil

INTERVENTIONS:
Other: 3% kanuka oil — To assess the efficacy in patients with mild atopic dermatitis, 3% kanuka oil will be applied twice a day for 28 days. 3% kanuka oil is a naturally occurring extract from the kanuka tree and is considered an over-the-counter agent.

SUMMARY:
Atopic dermatitis is a common disease affecting millions worldwide. A common associated symptom in this population is pruritus. We seek to investigate the use of an natural, over-the-counter cosmeceutical to help this population

DETAILED DESCRIPTION:
There are many treatment options available for atopic dermatitis yet many patients still suffer from the underlying symptomatology. It is important to explore other treatment alternatives to help this population.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 12 years, diagnosis of atopic dermatitis for longer than 2 years, investigator's static global assessment score of either 2 or 3, and initial worst itch numerical rating scale (WI-NRS) for itch greater than 4.

Exclusion Criteria:

* the use of topical or systemic corticosteroids within 28 days of entering the study, the use of any other non-emollient therapy within 28 days of entering the study,nursing, and pregnancy

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
ISGA | 28 days
  Investigator scale to determine imporvement in condition
WI-NRS | 28 days
  Scale generated by patient's responses to survey questions to assess improvement in itch

CONTACTS AND LOCATIONS:
Locations (1):
- Berlin Center, Boynton Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No
The individual participant data will be confidential and not shared unless authorized by the participant

REFERENCES:
- [Background] Shortt N, Martin A, Kerse K, Shortt G, Vakalalabure I, Barker L, Singer J, Black B, Liu A, Eathorne A, Weatherall M, Rademaker M, Armour M, Beasley R, Semprini A; Medical Research Institute of New Zealand's Pharmacy Research Network. Efficacy of a 3% Kanuka oil cream for the treatment of moderate-to-severe eczema: A single blind randomised vehicle-controlled trial. EClinicalMedicine. 2022 Jul 15;51:101561. doi: 10.1016/j.eclinm.2022.101561. eCollection 2022 Sep. PMID 35865740